CLINICAL TRIAL: NCT04846517
Title: Multilocus Repetitive Transcranial Magnetic Stimulation for Anorexia Nervosa (MULTI-REX): A 4-week Open-Trial Pilot Study
Brief Title: rTMS for Aneroxia Nervosa in Youth
Acronym: MULTI-REX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Assistant Professor- UCLA Neuromodulation Division, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-001905
Record Dates: First submitted 2021-03-12; First posted 2021-04-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Anorexia Nervosa
Keywords: AN; TMS
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMS Treatment (Other): iTBS treatment: Trains of 50 Hz pulses every 200 ms lasting 2 s, with an 8 s intertrain interval (ITI), repeated 60 times 1800 total pulses each day Treatment Duration: 9 minutes Location: Left DLPFC LF-rTMS treatment: Delivered immediately after iTBS treatment as described above.
  SMA will involve a continuous train of 1 Hz stimulation for a total of 1200 pulses lasting 20 minutes Treatment Duration: 20 minutes Location: SMA
  Interventions: Device: Transcranial Magnetic Treatment

INTERVENTIONS:
Device: Transcranial Magnetic Treatment — iTBS treatment: Trains of 50 Hz pulses every 200 ms lasting 2 s, with an 8 s intertrain interval (ITI), repeated 60 times 1800 total pulses each day Treatment Duration: 9 minutes Location: Left DLPFC
  LF-rTMS treatment: Delivered immediately after iTBS treatment as described above.
  SMA will involve a continuous train of 1 Hz stimulation for a total of 1200 pulses lasting 20 minutes Treatment Duration: 20 minutes Location: SMA

SUMMARY:
This study will examine the feasibility of off-label multilocus repetitive transcranial magnetic stimulation (rTMS) for symptoms of Anorexia Nervosa in participants between the ages of 14-24. rTMS is a non-invasive, brain-based intervention that uses magnets to deliver energy to the brain. The investigators will also see if patients receiving multilocus rTMS show any improvements in their eating disorder, mood, anxiety, and obsessions and compulsions (if present). Participants will receive daily intervention with off-label multilocus rTMS for 20 total treatments. Participants will also be asked to complete mental health and well-being surveys, physical measurements, and 2 brain imagining scans (MRIs) at baseline, and at study end. The investigators will also ask participants to complete surveys are 1-month and 3-months after the final rTMS session. The target enrollment for this study is 45 participants.

ELIGIBILITY:
Inclusion Criteria:

1. youth aged 14-24 with DSM-5 AN-restricting (ANR) or AN-binge-eating-purging (ANBP) type as determined by the MINI-KID/MINI and clinical interview;
2. YBC-EDS score≥16,
3. baseline CGI-S score ≥4,
4. English speaking (as this complement of questionnaires are available in English)
5. on stable psychotropic medication (if any) for the preceding 4 weeks (i.e., SSRIs, atypical antipsychotics and benzodiazepines of doses <1 mg lorazepam equivalent daily),
6. medically stable, as determined by their treating clinician, and
7. not deemed to be at high risk of imminent suicidal behavior by initial study psychiatrist assessment and referring provider/team, and no endorsement of items 4 or 5 on the Severity of Ideation Subscale of the C-SSRS.
8. For women: not currently pregnant and on reliable birth control if sexually active (as the effects of rTMS on the unborn fetus are unknown).

Exclusion Criteria:

1. a lifetime history of psychosis, mania, or seizure disorder
2. active suicidality as determined by clinical assessment by MD or PhD, and endorsement of items 4 or 5 on the Severity of Ideation Subscale of the C-SSRS.
3. unstable neurological disorder,
4. metal in head/eye,
5. inability to tolerate MRI,
6. at high risk of alcohol withdrawal or substance intoxication,
7. diagnosis of pervasive development disorder,
8. medical instability as determined by primary care provider and/or referring clinician (i.e., unstable electrolytes in the setting of worsening binge-eating/purging, cardiac arrhythmias requiring Holter or other intensive monitoring),
9. For women: pregnant or not using a reliable form of birth control.

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown-Cornell Eating Disorder Scale (YBC-EDS) | through study completion, an average of 6 weeks
  The YBC-EDS consists of a 65-item symptom checklist, followed by 19 questions. Although the thoughts and behaviors included in the YBC-EDS symptom checklist are fairly extensive, patients may add any eating-related thoughts or behaviors that are not part of the checklist. Once the preoccupations and rituals checklists have been completed, four core questions are then asked regarding preoccupations and four regarding rituals, yielding a Preoccupations Subtotal, Rituals Subtotal, and a YBC-EDS Total Score. A provisional score assessing the patient's motivation for change can also be calculated, and has shown to be an important predictor of treatment outcome. The YBC-EDS Interview takes between 45-60 minutes to administer.

IPD SHARING:
Plan to Share IPD: No